CLINICAL TRIAL: NCT03921658
Title: The Role of Cytomegalovirus and Inflammation on Patient Symptoms and Outcomes in Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2019NTLS030
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples at up to 3 time points
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 - Cross-sectional (within 2 years of diagnosis): Individuals diagnosed and treated for ovarian cancer in past two years, will complete 1 study measure
- Cohort 2- Prospective (from diagnosis): Individuals newly diagnosed with ovarian cancer, will complete 3 study measures (baseline/diagnosis, completion of chemotherapy, one year post-diagnosis)

SUMMARY:
Cytomegalovirus (CMV), a widely prevalent virus in the general US population, has been shown to be associated with increased inflammation and mortality. Previous small pilot studies have demonstrated that latent CMV may be reactivated during chemotherapy in cancer patients, and may be associated with unfavorable cancer outcomes such as fatigue and increased mortality.

The central research idea for this study, supported by previous preliminary data, is that CMV reactivation is an unrecognized complicating factor in the treatment of ovarian cancer that impacts patient outcomes. The overarching goals of this observational study are:

* To assess how CMV infection is associated with ovarian cancer symptoms over the course of the disease and its treatment.
* To describe the relationship between CMV reactivation in ovarian cancer patients, survival, fatigue, and other QOL outcomes, both cross-sectionally and longitudinally.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Ability to read and write in English
* women with newly diagnosed with ovarian, primary peritoneal, or fallopian tube cancer
* Treatment plan includes chemotherapy
* Able to provide written voluntary consent before performance of any study related procedure.
* Cohort 1 only: within 2 years of completing initial chemotherapy treatment
* Cohort 2 only: prior to starting chemotherapy

Exclusion Criteria:

* Inability to provide informed written consent
* Previous exposure to chemotherapy
* Life expectancy < 3 months or in hospice care or nursing home

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed and/or treated for ovarian/Fallopian tube/primary peritoneal cancer by physicians in the Gynecologic Oncology Clinic at the University of Minnesota
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Cohort 1 - Cancer-related fatigue | post treatment
  Cancer-related fatigue will be measured using the Fatigue Symptom Inventory. The scale is composed of 14 items (one is not scored). A total Disruption Index is calculated by summing items 5-11 (each item ranges from 0-10). A lower score indicates lower fatigue. Possible range is 0-70.
Cohort 2 - Recurrence-free survival | 3 years
  Time from diagnosis to first known recurrence or death, censored at least follow-up if recurrence free and alive

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No